CLINICAL TRIAL: NCT02478242
Title: Trial to Assess the Efficacy and Safety of Nafamostat Mesilate During Continuous Renal Replacement Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Chan-Duck Kim, M.D., Ph.D., Associate Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUH_08-0023
Record Dates: First submitted 2015-06-11; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — nafamostat; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nafamostat mesilate group (Active Comparator): Nafamostat mesilate was used for maintenance anticoagulation during continuous renal replacement therapy.
  Interventions: Drug: Nafamostat mesilate
- No anticoagulation group (Placebo Comparator): Normal saline was used for maintenance anticoagulation during continuous renal replacement therapy.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Nafamostat mesilate — nafamostat mesilate use for anticoagulation
  Other Names: Futhan
  Arms: Nafamostat mesilate group
Drug: Normal saline
  Arms: No anticoagulation group

SUMMARY:
Randomized study to evaluate the efficacy and safety of nafamostat mesilate use during continuous renal replacement therapy in acute kidney injury patients at a high risk of bleeding.

DETAILED DESCRIPTION:
Patients were randomly assigned to the nafamostat mesilate (NM) group or the no anticoagulant (NA) group. In patients assigned to the NM group, NM (20mg/h) was used for maintenance anticoagulation. Whereas, in patients assigned to the NA group, normal saline (2mL/h) was infused for continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were admitted to the intensive care unit and required CRRT

  1. active bleeding such as gastrointestinal bleeding and intracranial hemorrhage,
  2. activated partial thromboplastin time > 60 s,
  3. prothrombin time-international normalized ratio > 2.0,
  4. thrombocytopenia (<100,000/µL), and
  5. surgery within 48 h before CRRT.

Exclusion Criteria:

* Pregnant or possibly pregnant women
* Patients who were allergic to nafamostat mesilate
* Patients who were hypercoagulable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of filters used per hour | 24 months

SECONDARY OUTCOMES:
Urea reduction ratio | 24 months
Survival rate | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Duck Kim, M.D., PhD, Principal Investigator — Associate Professor

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078